CLINICAL TRIAL: NCT01359774
Title: 31Phosphorus-Magnetic Resonance Spectroscopy and Huntington Disease
Brief Title: 31P-MRS and Huntington Disease
Acronym: PRO-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C10-56; 2011-A00137-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2012-09

CONDITIONS: Huntington Disease
Keywords: Energy; Metabolism; Spectroscopy
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Other)
  Interventions: Other: 31P-MR spectroscopy
- Huntington patients (Other)
  Interventions: Other: 31P-RMN spectroscopy

INTERVENTIONS:
Other: 31P-MR spectroscopy — Brain energy deficit is quantified using 31P-MR spectroscopy
  Arms: Healthy volunteers
Other: 31P-RMN spectroscopy — Brain energy deficit is quantified using 31P-RMN spectroscopy
  Arms: Huntington patients

SUMMARY:
The purpose of this study is to identify and quantify a brain energy deficit in Huntington patients, using 31P-RMN spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* 5<UHDRS<50
* Age>18 years
* Ability to undergo MR scanning
* Covered by french social security

Exclusion Criteria:

* Evidence of psychiatric disorder
* Attendant neurological disorder
* Contraindications to MRI (claustrophobia, metallic or material implants)
* Severe head injury
* Unable to understand the protocol
* Pregnancy
* Failure to give informed consent
* Subjects with exclusion criteria required by french law (e.g. subjects who require a legally authorized representative to obtain consent)
* Unwillingness to be informed in case of abnormal MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Brain energy deficit in Huntington patients | one year
  31P-MRS allows quantification of high-energy phosphate metabolites such as ATP and phosphocreatine.
  Objective: to look at brain energy metabolism during rest and activation.

SECONDARY OUTCOMES:
Correlating a brain energy deficit with (i) biochemical parameters and (ii) clinical parameters in Huntington patients | one year
  Biochemical parameters include metabolites that we previously showed to be biomarkers in HD: branched chain amino acids and IGF1.
  Clinical parameters include UHDRS and TFC.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Mochel, MD, PhD, Principal Investigator — INSERM UMR S975 Institut du Cerveau et de la Moelle, AP-HP Département de Génétique, Université Pierre et Marie Curie, Paris France
Locations (1):
- Hopital de la Pitié-Salpetrière, Paris, France

REFERENCES:
- [Background] Mochel F, N'Guyen TM, Deelchand D, Rinaldi D, Valabregue R, Wary C, Carlier PG, Durr A, Henry PG. Abnormal response to cortical activation in early stages of Huntington disease. Mov Disord. 2012 Jun;27(7):907-10. doi: 10.1002/mds.25009. Epub 2012 Apr 19. PMID 22517114
- [Background] Mochel F, Haller RG. Energy deficit in Huntington disease: why it matters. J Clin Invest. 2011 Feb;121(2):493-9. doi: 10.1172/JCI45691. Epub 2011 Feb 1. PMID 21285522
- [Background] Mochel F, Charles P, Seguin F, Barritault J, Coussieu C, Perin L, Le Bouc Y, Gervais C, Carcelain G, Vassault A, Feingold J, Rabier D, Durr A. Early energy deficit in Huntington disease: identification of a plasma biomarker traceable during disease progression. PLoS One. 2007 Jul 25;2(7):e647. doi: 10.1371/journal.pone.0000647. PMID 17653274
- [Background] Mochel F, Benaich S, Rabier D, Durr A. Validation of plasma branched chain amino acids as biomarkers in Huntington disease. Arch Neurol. 2011 Feb;68(2):265-7. doi: 10.1001/archneurol.2010.358. No abstract available. PMID 21320997
- See also: European Huntington's Disease Network — http://www.euro-hd.net